CLINICAL TRIAL: NCT01984957
Title: Differential Study of Muscle Transcriptome in Patients With Neuromuscular Disease and Control Subjects
Brief Title: Differential Study of Muscle Transcriptome
Acronym: TRANE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Direction Générale de l'Offre de Soins (Other Government); Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: P110401
Record Dates: First submitted 2013-06-27; First posted 2013-11-15 (Estimated); Last update posted 2015-03-23 (Estimated); Status verified 2014-06

CONDITIONS: ALS; SMA; SBMA
Keywords: ALS; Motor neuron diseases; Transcriptome
MeSH Terms: conditions — Motor Neuron Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- disease (ALS, SMA or SBMA) (Other): muscle biopsy
  Interventions: Procedure: Muscle biopsy

INTERVENTIONS:
Procedure: Muscle biopsy — open muscular biopsy of the deltoid under local anaesthesia

SUMMARY:
To isolate biomarkers of ALS in muscle

DETAILED DESCRIPTION:
At present, there is no validated biological diagnostic marker for amyotrophic lateral sclerosis (ALS). The main objective of the study is to isolate a set of genes that are specifically dysregulated in muscle from ALS patients.

Gene profiling in muscle will be compared between ALS patients and patients with other motor neuron diseases (SMA and SBMA)

ELIGIBILITY:
Inclusion criteria :

- Patient with ALS, SMA, or SBMA

Exclusion criteria :

* Indication against biopsy (allergy to anesthetics local haemostasis disorders)
* Treatments that can affect muscle metabolism

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2013-01; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Gene expression levels | day 1
  Gene expression levels in muscle as determined By microarrays (transcriptome analysis)

SECONDARY OUTCOMES:
muscle denervation | day 1
  Severity of muscle denervation as determined by histological analysis of muscle
Functional evaluation | day 1
  ALSFRS-R, Manual Muscle Testing and Slow Vital Capacity

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-Francois Pradat, MD, PhD, Principal Investigator — APHP
Locations (1):
- Centre d'évaluation Thérapeutique, Dr LACOMBLEZ, Paris, France